CLINICAL TRIAL: NCT00512655
Title: Randomized Controlled Trial to Reduce Falls Incidence Rate in Frail Elderly
Brief Title: Trial to Reduce Falls Incidence Rate in Frail Elderly
Acronym: CP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Extremely difficult recruitment. Preliminary analysis showed no effect of the intervention.
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Stichting Nuts Ohra (Other)
Responsible Party: Prof. Dr. MGM Olde Rikkert, Radboud University Nijmegen Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CP MM 19-08-12-05-30-08; SNO-T-0601-60; ZonMw 920-03-457
Record Dates: First submitted 2007-08-07; First posted 2007-08-08 (Estimated); Last update posted 2010-07-07 (Estimated); Status verified 2010-06

CONDITIONS: Accidental Falls
Keywords: Fear of falling; Intraindividual variability; Cognition; Fall prevention; Fear; Frail elderly; Intervention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Intervention: 5 week training program, 2 sessions per week (total of 10 sessions). Training includes both the patient and the caregiver. The training consists of two components: a cognitive and a physical component.
  Interventions: Behavioral: Fall prevention course
- 2 (No Intervention): Usual care.

INTERVENTIONS:
Behavioral: Fall prevention course — Duration: 5 weeks, 2 sessions of 2 hours per week: 10 sessions in total.
  Arms: 1

SUMMARY:
Background: Approximately 750,000 elderly Dutch people fall at least once a year, which often results in physical injuries and a fear of falling, with high costs and far-reaching consequences on functionality, physical activity, quality of life and mental well-being. Falling is not only a burden for patients, it is also a burden for their caregivers. Recurrent falling is a complex problem. However, the pathophysiological background of falls, gait problems and dementia is largely unknown. The general pathophysiological hallmark of aging is a liability in homeostatic mechanisms of organs. This liability results in an impaired ability to adapt to stress and in increased biological variation in outcome measures within individuals. In this study the investigators aim at developing an intervention to reduce recurrent falling in frail elderly fallers.

Hypotheses: The investigators hypothesize that the intervention program will decrease the number of falls and fear of falling and increase mental well-being, physical activity and functional performance in frail elderly people with a history of recurrent falling. In addition, the burden on the caregivers will be reduced due to the intervention and will be cost-effective. Furthermore, the investigators hypothesize that patients with a high short-term intra-individual biological variability in gait and cognition variables have a higher risk of falling, worse gait performance and cognitive decline after long term follow-up.

Study Design: Randomized, controlled, single-blind trial.

Study Population: 160 patients referred to a geriatric outpatient clinic, who fell at least once in the last 6 months and their primary caregivers (N=160).

Intervention: A multifaceted fall prevention program for frail elders to reduce falls incidence rate, consisting of physical and cognitive components. Moreover, it includes a training program for caregivers in which they learn to support and give advice to the patients, aiming to decrease the burden on the caregivers.

Primary Outcome Measures: The fall incidence rate is the primary outcome measure. Total observation time of falls will be 6 months after the start of the intervention.

Secondary Outcome Measures: In the patients, the secondary outcome measures are fear of falling (FES), quality of life (MOS-20), depression and general anxiety, functional performance in activities of daily living, physical activity, mobility, gait parameters, body sway and biomarkers of endothelial function and frailty. For the caregiver, the secondary outcome measures are caregiver's burden, mood and quality of life. In addition, intraindividual variability of cognition, balance and gait in both patients and caregivers, will be assessed and cost-effectiveness of the intervention will also be determined.

DETAILED DESCRIPTION:
Nature and Extent of the Burden and Risks Associated with Participation, Benefit and Group Relatedness: The outcome of this study may have important reflections on protocols to prevent falling among elders and on health care decision makers to stimulate starting new fall clinics and implement these protocols. Through this study, the well-being and functionality of frail elders and their caregivers could be improved. As falling has an enormous economic burden, a new effective fall prevention intervention could reduce health care costs substantially. The tests consisting of questionnaires and gait and balance measurement are non-invasive and safe. Taking blood samples is an invasive procedure, although no serious adverse effects are expected. There are no foreseeable risks associated with participation in this study. However, a burden will be placed on participating individuals because the training sessions and measurements are time-consuming.

ELIGIBILITY:
Inclusion Criteria:

* At least one fall in the last 6 months
* Living in their own home or in a home for the aged
* Availability of a primary caregiver caring for the patient at least once a week
* Ability to walk 15 meters independently (use of a walking aid is permitted)
* Life expectancy of more than 6 months, as judged by their geriatrician

Exclusion Criteria:

* Dyads of patients and caregivers in whom outcome assessment is highly unlikely to succeed, for example because they proved not to be able to register falls in the three months before randomization, will be excluded
* MMSE score of less than 15
* On the waiting list for a nursing home

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2008-01; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Falls incidence rate | 6 months

SECONDARY OUTCOMES:
Burden for the caregiver | 4 measurements within 6 months
Quality of life (MOS-20) | 4 measurements within 6 months
Balance confidence | 4 measurements within 6 months
Depression and general anxiety | 4 measurements within 6 months
Functional performance and activities of daily living | 4 measurements within 6 months
Mood | 4 measurements within 6 months
Physical activity | 4 measurements within 6 months
Mobility | 4 measurements within 6 months
Balance | 4 measurements within 6 months
Cognition | 4 measurements within 6 months
Fear of falling (FES) | 4 measurements within 6 months
Mental well being | 4 measurements within 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. M. Olde Rikkert, MD PhD, Principal Investigator — Radboud University Medical Center
Locations (3):
- Netherlands (3):
  - Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland
  - Rijnstate Ziekenhuis, Arnhem
  - CWZ, Nijmegen

REFERENCES:
- [Derived] Faes MC, Reelick MF, Melis RJ, Borm GF, Esselink RA, Rikkert MG. Multifactorial fall prevention for pairs of frail community-dwelling older fallers and their informal caregivers: a dead end for complex interventions in the frailest fallers. J Am Med Dir Assoc. 2011 Jul;12(6):451-8. doi: 10.1016/j.jamda.2010.11.006. Epub 2010 Dec 24. PMID 21450224